CLINICAL TRIAL: NCT06399315
Title: A Randomised, Double-Blind, Placebo-Controlled, First-in-Human Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Ascending Doses of ZE46-0134 in Healthy Volunteers
Brief Title: Study of Single and Multiple Ascending Doses of ZE46-0134 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lomond Therapeutics Holdings, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ZE46-0134-0001; CT-2023-CTN-03208-1 (Other: therapeutic goods administration)
Record Dates: First submitted 2024-05-01; First posted 2024-05-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: AML
MeSH Terms: interventions — Rabeprazole; Itraconazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-Blind, Placebo-Controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Level 1 Single dose (Experimental): Dose level 1. SAD study part. 6 participants will receive the study drug and 2 participants will receive placebo
  Interventions: Drug: ZE46-0134 or placebo
- Level 2 Single dose (Experimental): Dose level 2. SAD study part. 6 participants will receive the study drug and 2 participants will receive placebo
  Interventions: Drug: ZE46-0134 or placebo
- Level 3 Single dose (Experimental): Dose level 3. SAD study part. 6 participants will receive the study drug and 2 participants will receive placebo
  Interventions: Drug: ZE46-0134 or placebo
- Level 2 Single dose after food (Experimental): Dose level 2 with a fat meal. SAD study part. 6 participants will receive the study drug and 2 participants will receive placebo
  Interventions: Drug: ZE46-0134 or placebo
- Level 4 Single dose (Experimental): Dose level 4. SAD study part. 6 participants will receive the study drug and 2 participants will receive placebo
  Interventions: Drug: ZE46-0134 or placebo
- Level 1 Multiple doses (Experimental): Dose level 1. MAD study part. 6 participants will receive the study drug and 2 participants will receive placebo
  Interventions: Drug: ZE46-0134 or placebo
- Level 1 Multiple doses + rabeprazole (Experimental): Dose level 2. MAD study part. 6 participants will receive the study drug and 2 participants will receive placebo. The drug is co-administered with rabeprazole
  Interventions: Drug: ZE46-0134 or placebo; Drug: Rabeprazole, 20mg oral
- Level 2 Multiple doses (Experimental): Dose level 2. MAD study part. 6 participants will receive the study drug and 2 participants will receive placebo
  Interventions: Drug: ZE46-0134 or placebo
- Level 3 Single dose with itraconazole (Experimental): Dose level 3. SAD study part. 6 participants will receive the study drug and 2 participants will receive placebo, in conjunction with itraconazole
  Interventions: Drug: ZE46-0134 or placebo; Drug: Itraconazole (200 mg)
- Level 5 Single dose (Experimental): Dose level 5. SAD study part. 6 participants will receive the study drug and 2 participants will receive placebo
  Interventions: Drug: ZE46-0134 or placebo
- Level 6 Single dose (Experimental): Dose level 6. SAD study part. 6 participants will receive the study drug and 2 participants will receive placebo
  Interventions: Drug: ZE46-0134 or placebo
- Level 3 Multiple doses (Experimental): Dose level 3. MAD study part. 6 participants will receive the study drug and 2 participants will receive placebo
  Interventions: Drug: ZE46-0134 or placebo
- Level 4 Multiple doses (Experimental): Dose level 4. MAD study part. 6 participants will receive the study drug and 2 participants will receive placebo
  Interventions: Drug: ZE46-0134 or placebo
- Level 5 Multiple doses (Experimental): Dose level 5. MAD study part. 6 participants will receive the study drug and 2 participants will receive placebo
  Interventions: Drug: ZE46-0134 or placebo

INTERVENTIONS:
Drug: ZE46-0134 or placebo — The patients will receive ZE46-0134 or placebo
  Other Names: lomonitininb
Drug: Rabeprazole, 20mg oral — Rabeprazole 20 mg daily will be administered for 2 prior ZE46-0134 and 7 co-administered
  Arms: Level 1 Multiple doses + rabeprazole
Drug: Itraconazole (200 mg) — Itraconazole 200 mg BID
  Arms: Level 3 Single dose with itraconazole

SUMMARY:
This is a clinical study aiming to assess pharmacokinetics and biomarker evidence of ZE46-0134 efficacy in Healthy Volunteers after single and multiple daily doses of the study drug

DETAILED DESCRIPTION:
This is a Phase 1, double-blind, placebo-controlled, dose escalation study to evaluate the safety, tolerability, PK, PD of orally administered ZE46-0134 in Healthy Volunteers. The study will be conducted in 2 parts: a single ascending dose (SAD) part at up to 6 dose levels and a multiple ascending dose (MAD) part at up to 5 dose levels. Evaluation of dose levels will be conducted in a sequential fashion with lower dose levels evaluated first in the sequence. Dosing in each cohort will start with two sentinel participants with one of the two sentinels randomised to receive ZE46-0134 and the other randomised to receive placebo. The food-effect will be investigated in SAD part and safety/PK of co-administration with rabeprazole will be investigated in MAD part.

ELIGIBILITY:
Inclusion Criteria:

* 1. Must have given written informed consent before any study-related activities are carried out and must be able to understand the full nature and purpose of the trial, including possible risks and adverse effects.

  2. Adult males and females, 18 to 55 years of age (inclusive) at screening. 3. Body mass index (BMI) ≥ 18.5 and ≤ 32.0 kg/m2, with a body weight (to 1 decimal place) ≥ 50.0 kg at screening.

  4. Medically healthy without clinically significant abnormalities (in the opinion of the Investigator) at the screening visit and prior to dosing

Exclusion Criteria:

1. History or presence of significant cardiovascular, pulmonary, hepatic, renal, haematological, gastrointestinal, endocrine, immunologic, dermatologic or neurological disease, including any acute illness or major surgery within the past 3 months determined by the PI to be clinically significant.
2. Acute infections within 4 weeks prior to screening or current infection that requires systemically absorbed antibiotic, antifungal, antiparasitic or antiviral medications.
3. Presence or history of any abnormality or illness, including gastrointestinal surgery, which in the opinion of the PI may affect absorption, distribution, metabolism or elimination of the study drug.
4. Any history of malignant disease in the last 5 years (excludes surgically resected skin squamous cell or basal cell carcinoma).
5. Any screening laboratory result outside the normal laboratory reference range (as confirmed upon repeated testing) and deemed clinically significant by the PI.
6. Presence of clinically relevant immunosuppression from, but not limited to, immunodeficiency conditions such as common variable hypogammaglobulinemia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 112 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-08-26 (Actual)

PRIMARY OUTCOMES:
Plasma concentration | 72 hours for SAD, 10 days for MAD
  Plasma concentration, ng/mL

SECONDARY OUTCOMES:
Incidence of AEs | 8 days in SAD part, 17 days for MAD part
  Incidence of Adverse Events observed during the study
Incidence of drug-related AEs | 8 days in SAD part, 17 days for MAD part
  Incidence of Adverse Events observed during the study deemed related to the study drug by the Investigator
Incidence of SAEs | 8 days in SAD part, 17 days for MAD part
  Incidence of Serious Adverse Events observed during the study
Incidence of lab deviations | Time Frame: 8 days in SAD part, 17 days for MAD part
  Incidence of clinically relevant deviations in the clinical laboratory parameters

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research Ltd, Perth, Nedlands, Australia